CLINICAL TRIAL: NCT00469781
Title: Bromfenac BID Plus Prednisolone Acetate BID Versus Bromfenac BID Plus Prednisolone QID for the Prevention of Cystoid Macular Edema and Retinal Thickening
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Center For Excellence In Eye Care (Other)
Responsible Party: Carlos Buznego, MD, The Center for Excellence in Eye Care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5306
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Cystoid Macular Edema,; Retinal Thickening
MeSH Terms: conditions — Macular Edema | interventions — bromfenac

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: 1. Pred Forte
- 2 (Other)
  Interventions: Drug: 2. Xibrom (Bromfenac)

INTERVENTIONS:
Drug: 2. Xibrom (Bromfenac) — Group 1 and 2: 1 drop(Instill one drop in the eye that was operated on twice daily)3 days prior to surgery and 4 doses during dilation immediately before the procedure. Use for 4 weeks after surgery.
  Arms: 2
Drug: 1. Pred Forte — Group 1 Instill one drop in the eye that was operated on four times a day starting on day of surgery and use for four weeks.
  Group 2 Instill one drop in the eye that was operated on twice a day starting on day of surgery and use for four weeks.
  Arms: 1

SUMMARY:
The objective of this study is to determine if twice-daily dosing of prednisolone (Pred Forte) is as effective as four-times-daily dosing of prednisolone for the prevention of retinal thickening and cystoid macular edema (CME) when either regimen is used concomitantly with twice-daily bromfenac.

ELIGIBILITY:
Inclusion Criteria:

* · Male or female > 18 years of age scheduled to undergo cataract surgery

  * Must be in good general health. Patients with systemic diseases will be enrolled only if there are no ocular manifestations of their disease (ie diabetics with normal retinal exams)
  * Expected visual outcome of 20/25 or better.
  * Ability to provide informed consent and likely to complete all study visits

Exclusion Criteria:

* · Known contraindication to any study medication or any of their components

  * Uncontrolled systemic disease
  * Required use of ocular medications other than the study medications during the study
  * Abnormal pre-operative OCTs
  * Diabetic patients with a history of macular edema or diabetic retinopathy
  * AMD, epi-retinal membranes, retinal vein occlusion, or any pre-existing macular disease
  * Only one eye of each patient can be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2007-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Cystoid Macular Edema | 11 months

SECONDARY OUTCOMES:
Retinal Thickening | 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Buznego, MD, Principal Investigator — The Center for Excellence in Eye Care
Locations (1):
- The Center for Excellence in Eye Care, Miami, Florida, United States